CLINICAL TRIAL: NCT02104778
Title: Effect of Dexamethasone and Epinephrine on the Duration of Sciatic Nerve Blocks With Ropivacaine in Ankle and Foot Surgery
Brief Title: Effect of Dexamethasone and Epinephrine on the Duration of Sciatic Nerve Blocks With Ropivacaine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Sangjin Park, assistant professor, Yeungnam University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: apsj20140401
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dexamethasone (Experimental): Dexamethasone 8 mg is added to 0.5% ropivacaine 20 ml for sciatic nerve block.
  Interventions: Drug: Dexamethasone
- Control (Placebo Comparator): Normal saline 1 ml is added to 0.5% ropivacaine 20 ml for sciatic nerve block.
- epinephrine (Experimental): Epinephrine 1:200,000 is added to 0.5% ropivacaine 20 ml for sciatic nerve block.
  Interventions: Drug: Epinephrine

INTERVENTIONS:
Drug: Dexamethasone — In dexamethasone group, dexamethasone 8 mg is added to 0.5% ropivacaine 20 ml for sciatic nerve block.
  Arms: Dexamethasone
Drug: Epinephrine — Epinephrine 1:200,000 is added to 0.5% ropivacaine 20 ml for sciatic nerve block
  Arms: epinephrine

SUMMARY:
The aim of the present study is to test that adding dexamethasone or epinephrine significantly prolongs the duration of sciatic nerve blocks with ropivacaine and that the magnitude of the effect differs among dexamethasone and epinehrine.

DETAILED DESCRIPTION:
In a double-blinded trial utilizing single-injection sciatic nerve block, patients are randomly assigned to one of three groups: control: 0.5% ropivacaine adding normal saline; epinephrine: 0.5% ropivacaine adding epinephrine; dexamethasone: 0.5% ropivacaine adding dexamethasone. We assess time to first analgesic request after post-anaesthesia care unit discharge.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I and II
* patients undergoing elective hallux valgus repair

Exclusion Criteria:

* patients receiving chronic analgesic therapy
* diabetes
* peripheral neuropathies
* psychiatric disorders
* hypersensitivity to amide local anesthetics
* renal disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
time to first analgesic request after postanesthetic care unit discharge | from arrival in postanesthetic care unit to 72 hours after operation
  A blinded observer interview patients at arrival in postanesthetic care unit, 6 hour, 24 hour, 48 hour, 72 hour after operation.

SECONDARY OUTCOMES:
time of recovery of motor and sensory functions on the operated foot | from arrival in postanesthetic care unit to 72 hours after operation
  The time of recovery of motor (ability to move the ankle) and sensory (recovery of normal pinprick sensation) functions on the operated foot is recorded by the blinded observer at arrival in postanesthetic care unit, 6 hour, 24 hour, 48 hour, 72 hour after operation.

CONTACTS AND LOCATIONS:
Overall Officials: Sangjin Park, M.D., Principal Investigator — Department of Anesthesiology and Pain Medicine, College of medicine, Yeungnam University, Daemyung-Dong, Nam-Gu, Daegu, Republic of Korea
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yeungnam University hospital, Daegu, South Korea